CLINICAL TRIAL: NCT01232296
Title: An Open-label, Randomized, Multi-center, Phase II Study to Compare the Safety and Efficacy of TKI258 Versus Sorafenib as First-line Treatment in Adult Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of Dovitinib Versus Sorafenib in Adult Patients With Hepatocellular Carcinoma (HCC) as a First Line Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2208
Record Dates: First submitted 2010-09-30; First posted 2010-11-02 (Estimated); Results first posted 2015-12-04 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; HCC; Liver cancer; Child Pugh A; HCC Stage C
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Sorafenib

ARMS (2):
- TKI258 (Experimental): capsule
  Interventions: Drug: dovitinib
- Sorafenib (Experimental): tablet
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: dovitinib — 500 mg p.o. o.d. 5 days on/2 days off
  Other Names: TKI258
  Arms: TKI258
Drug: sorafenib — 400 mg p.o. b.i.d.
  Arms: Sorafenib

SUMMARY:
The purpose of this open-label, randomized, phase II study is to compare the safety and efficacy of dovitinib versus sorafenib as first-line treatment in adult patients with advanced Hepatocellular Carcinoma (HCC). This trial will be opened in countries of the Asia-Pacific region.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of advanced Hepatocellular Carcinoma (HCC) according to the AASLD Guidelines

* Advance HCC Stage B and C according to BCLC staging classification
* Child Pugh A
* At least one measurable lesion as assessed by CT or MRI
* ECOG PS of 0 or 1
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Prior systemic therapy for HCC
* Brain metastases
* Active bleeding (including variceal bleeding as the result of esophageal varices) Patients who have received a liver transplant or are awaiting an immediate transplant

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- China (4):
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
- Hong Kong (2):
  - Novartis Investigative Site, Shatin, New Territories, Hong Kong
  - Novartis Investigative Site, Hong Kong
- Japan (3):
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sayama, Osaka
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (4):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
- Thailand (4):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
  - Novartis Investigative Site, Khon Kaen
  - Novartis Investigative Site, Songkhla

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 165 Participants were screened and randomized. However 3 participants discontinued prior to recieving study drug. The number enrolled in the protocol section reflects the randomized participants who received study drug.
Groups:
- TKI258: 500 mg capsules p.o. o.d. 5 days on/2 days off
- Sorafenib: 400 mg tablet p.o. b.i.d.
Period: Overall Study
Arm/Group | TKI258 | Sorafenib
Started | 82 | 83
Full Analysis Set | 82 | 83
Safety Set | 79 (The Safety Set includes all patients who received at least one dose of study medication) | 83
Completed | 0 | 0
Not Completed | 82 | 83
Not completed — Adverse Event | 24 | 12
Not completed — Physician Decision | 1 | 1
Not completed — Progressive disease | 43 | 61
Not completed — Study terminated by sponsor | 0 | 1
Not completed — Technical problems | 3 | 0
Not completed — Subject/guardian decision | 10 | 2
Not completed — Death | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TKI258 | Sorafenib | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (12.16) | 56.2 (11.72) | 55.8 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 73 | 67 | 140

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival - Overall Survival
Description: The overall survival (OS), defined as the time from date of randomization to the date of death from any cause. If a patient was not known to have died at the date of analysis cut-off, OS was censored at the last date of contact. Survival information was collected every 6 wks until at least 130 deaths have been observed
Time Frame: Every 6 weeks from date of randomization until the patient has progressed, or the patient can no longer be followed, or at least 130 deaths have been observed in the study, whichever came first.
Population: The Full Analysis Set (FAS) comprises of all patients to whom study treatment had been assigned by randomization. According to the intent to treat principle, patients were analyzed according to the treatment (and strata) they were assigned to during the randomization procedure.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | TKI258 | Sorafenib
Number analyzed (Participants) | 82 | 83
Weeks | 33 [25.7 to 39] | 39.4 [22.6 to 56.1]

2. Secondary Outcome: Time to Tumor Progression (Tumor Assessment)
Description: Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1). For target lesions, disease progression mean at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. For non-target lesions, disease progression refers to unequivocal progression of existing non-target lesions. In addition, the appearance of new lesions is always considered as disease progression.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | TKI258 | Sorafenib
Number analyzed (Participants) | 82 | 83
Weeks | 17.6 [12.3 to 18.4] | 17.9 [12.3 to 18.9]

3. Secondary Outcome: Disease Control Rate (Tumor Assessment)
Description: Disease Control Rate (DCR) is defined as the proportion of patients whose best overall response is either complete response [CR], partial response [PR] or stable disease [SD] according to RECIST 1.1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TKI258 | Sorafenib
Number analyzed (Participants) | 82 | 83
Participants
  Complete response (CR) | 0 | 1
  Partial response (PR) | 5 | 8
  Stable disease (SD) | 42 | 44
  Progressive disease | 17 | 22
  Unknown (UNK) | 18 | 8

4. Secondary Outcome: Time to Definitive Deterioration in ECOG Performance Status (PS)
Description: Time to definitive deterioration on ECOG PS scale (by at least one point) was defined as the time from the date of randomization to the date of definitive deterioration of the ECOG PS by at least one category of the score from baseline or to the date of death whichever occurred earlier. 0 is Fully active, able to carry on all pre-disease performance without restriction, 1 is Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work and 2 is ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
Time Frame: as for outcome 1
Population: The Full Analysis Set (FAS): all patients to whom study treatment had been assigned by randomization. According to the intent to treat principle, patients were analyzed according to the treatment (and strata) they were assigned to during the randomization procedure. Only Total number of definitive deterioration events included in the analysis
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | TKI258 | Sorafenib
Number analyzed (Participants) | 82 | 83
Weeks | 22.3 [12.6 to 34.0] | 21.3 [13.6 to NA] — NA -The upper bound of the 95% CI is not estimable because of the high censoring proportion (43 censored patients out of 83 patients, or 51.8%).

5. Secondary Outcome: Pharmacokinetic (PK) Parameter of Cmax Following a Single Dose of TKI258
Description: Cmax will be evaluated after a single dose of TKI258 following a 5 days on/2 days off dosing schedule. Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after a single dose administration (mass x volume - 1).
Time Frame: Week 1 day 1, week 4 day 5
Population: The Full-PK analysis set: all patients who were selected for full PK sampling and provided at least one evaluable PK concentration profile
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | TKI258
Number analyzed (Participants) | 71
(ng/mL)
  Week 1 Day 1 (n=71) | 326.25 (100.405)
  Week 4 Day 5 (n=23) | 364.04 (131.973)

6. Secondary Outcome: Pharmacokinetic (PK) Parameter of Tmax Following a Single Dose of TKI258
Description: Tmax will be evaluated after a single dose of TKI258 following a 5 days on/2 days off dosing schedule. Tmax is the time to to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after a single dose administration (time)
Time Frame: Week 1 day 1, week 4 day 5
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | TKI258
Number analyzed (Participants) | 71
hours
  Week 1 Day 1(71) | 6 (NA) [3 to 24]
  Week 4 Day 5 (n=23) | 5.9 (NA) [0.0 to 6.1]

7. Secondary Outcome: Pharmacokinetic (PK) Parameter of AUCtau Following a Single Dose of TKI258
Description: The mean AUC from time zero to the last measurable concentration sampling time (t last) (mass x time x volume-1)
Time Frame: Week 1 day 1, week 4 day 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: (ng.h/mL)
Arm/Group | TKI258
Number analyzed (Participants) | 71
(ng.h/mL)
  Week 1 Day 1 | 5774.69 (1616.159)
  Week 4 Day 5 (n=23) | 6493.99 (2409.119)

ADVERSE EVENTS:
Arm/Group | TKI258 | Sorafenib
Serious Adverse Events (participants affected / at risk) | 40/79 | 34/83
Other Adverse Events (participants affected / at risk) | 77/79 | 80/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TKI258 (N=79) | Sorafenib (N=83)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2
ASCITES (Gastrointestinal disorders) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 3
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 1
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 2
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 2
VOMITING (Gastrointestinal disorders) | 2 | 1
FATIGUE (General disorders) | 3 | 1
OEDEMA PERIPHERAL (General disorders) | 2 | 0
PYREXIA (General disorders) | 10 | 5
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
HEPATIC FUNCTION ABNORMAL (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 0
LIVER ABSCESS (Infections and infestations) | 0 | 1
PERITONITIS BACTERIAL (Infections and infestations) | 0 | 2
SEPSIS (Infections and infestations) | 1 | 2
SEPTIC SHOCK (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 3 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 3 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
HEPATOCELLULAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LIVER CARCINOMA RUPTURED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 2 | 0
HEADACHE (Nervous system disorders) | 1 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 3 | 2
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 0
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 1 | 0
AORTIC DISSECTION RUPTURE (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 1
HYPERTENSION (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TKI258 (N=79) | Sorafenib (N=83)
ANAEMIA (Blood and lymphatic system disorders) | 10 | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 | 2
TINNITUS (Ear and labyrinth disorders) | 5 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 7 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 | 16
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 | 11
ASCITES (Gastrointestinal disorders) | 10 | 7
CHEILITIS (Gastrointestinal disorders) | 4 | 0
CONSTIPATION (Gastrointestinal disorders) | 16 | 12
DIARRHOEA (Gastrointestinal disorders) | 48 | 35
DRY MOUTH (Gastrointestinal disorders) | 3 | 5
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 4 | 1
NAUSEA (Gastrointestinal disorders) | 32 | 16
STOMATITIS (Gastrointestinal disorders) | 13 | 11
VOMITING (Gastrointestinal disorders) | 31 | 10
FATIGUE (General disorders) | 27 | 13
MALAISE (General disorders) | 5 | 5
OEDEMA PERIPHERAL (General disorders) | 13 | 11
PYREXIA (General disorders) | 16 | 18
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 6 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 3
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 17 | 17
AMMONIA INCREASED (Investigations) | 4 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 23 | 21
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 | 3
BLOOD BILIRUBIN INCREASED (Investigations) | 20 | 19
BLOOD CREATININE INCREASED (Investigations) | 5 | 2
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 7 | 4
NEUTROPHIL COUNT DECREASED (Investigations) | 12 | 2
PLATELET COUNT DECREASED (Investigations) | 14 | 8
WEIGHT DECREASED (Investigations) | 19 | 17
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 7 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 31 | 24
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 | 5
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 10 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 2
DIZZINESS (Nervous system disorders) | 9 | 2
HEADACHE (Nervous system disorders) | 11 | 4
INSOMNIA (Psychiatric disorders) | 17 | 9
COUGH (Respiratory, thoracic and mediastinal disorders) | 13 | 8
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 7 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 | 8
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 5 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 4
ACNE (Skin and subcutaneous tissue disorders) | 9 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 19
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 7 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 4 | 2
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 11 | 55
PRURITUS (Skin and subcutaneous tissue disorders) | 8 | 5
RASH (Skin and subcutaneous tissue disorders) | 27 | 18
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 4 | 0
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 4 | 0
HYPERTENSION (Vascular disorders) | 17 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety